CLINICAL TRIAL: NCT07225647
Title: An Open-Label, Randomized, Two-part Study in Healthy Participants to Assess the Food Effect on the Pharmacokinetics of Admilparant To-Be-Marketed Tablet Formulations
Brief Title: A Study to Assess the Effect of Food on the Drug Levels of Admilparant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1052
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Treatment A (Experimental)
  Interventions: Drug: Admilparant
- Part 1: Treatment B (Experimental)
  Interventions: Drug: Admilparant
- Part 2: Treatment C (Experimental)
  Interventions: Drug: Admilparant
- Part 2: Treatment D (Experimental)
  Interventions: Drug: Admilparant

INTERVENTIONS:
Drug: Admilparant — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the effect of food on the drug levels of Admilparant

ELIGIBILITY:
Inclusion Criteria

* Participants must have a body mass index (BMI) of 18.0 kg/m2 to 32.0 kg/m2, inclusive, at screening.
* Participants must have a body weight of ≥ 50 kg for males and ≥ 45 kg for females at screening.

Exclusion Criteria

* Participants must not have any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
* Participants must not have had any previous exposure to Admilparant.
* Participants must not have a history of any severe drug allergy or drug reaction (such as anaphylaxis or hepatotoxicity).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 13 days
Area under the concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to 13 days
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to 13 days

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 13 days
Terminal half-life (T-HALF) | Up to 13 days
Apparent total body clearance (CLT/F) | Up to 13 days
Apparent volume of distribution (Vz/F) | Up to 13 days
Number of participants with adverse events (AEs) | Up to 13 days
Number of participants with a change in clinical laboratory values | Up to 13 days
Number of participants with a change in vital sign measurements | Up to 13 days
Number of participants with a change in physical examination results | Up to 13 days
Number of participants with a change in 12-lead electrocardiogram (ECG) results | Up to 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0002, Lenexa, Kansas
  - Local Institution - 0001, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com